CLINICAL TRIAL: NCT00691717
Title: A Study of the Safety and IOP-Lowering Efficacy of Anecortave Acetate in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Anecortave Acetate Safety in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-07-36
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Open-angle Glaucoma; Oular Hypertension
Keywords: Anecortave acetate; Open-angle glaucoma; IOP; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 24 mg Anecortave Acetate (Experimental): Anecortave Acetate Sterile Suspension, 30 mg/mL, single depot administration of 0.8 mL in the study eye
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- 48 mg Anecortave Acetate (Experimental): Anecortave Acetate Sterile Suspension, 60 mg/mL, single depot administration of 0.8 mL in the study eye
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL
- 60 mg Anecortave Acetate (Experimental): Anecortave Acetate Sterile Suspension, 75 mg/mL, single depot administration of 0.8 mL in the study eye
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 75 mg/mL
- Anecortave Acetate Vehicle (Placebo Comparator): Single depot administration of 0.8 mL in the study eye
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL — Single administration by anterior juxtascleral depot
  Arms: 24 mg Anecortave Acetate
Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL — Single administration by anterior juxtascleral depot
  Arms: 48 mg Anecortave Acetate
Drug: Anecortave Acetate Sterile Suspension, 75 mg/mL — Single administration by anterior juxtascleral depot
  Arms: 60 mg Anecortave Acetate
Other: Anecortave Acetate Vehicle — Single administration by anterior juxtascleral depot
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study was to evaluate the safety and intraocular-lowering efficacy of anecortave acetate depot when administered by anterior juxtascleral depot (AJD) for the treatment of elevated intraocular pressure (IOP) in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older with open-angle glaucoma (with or without pigment dispersion or pseudoexfoliation) or ocular hypertension.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patients with any form of glaucoma other than open-angle.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure at 8 am | Up to 6 months

SECONDARY OUTCOMES:
Percent of Patients Who Remained Rescue Medication-Free at Month 3 (8 am) | Month 3, 8 am

CONTACTS AND LOCATIONS:
Locations (1):
- Charleston, Charleston, South Carolina, United States